CLINICAL TRIAL: NCT05192239
Title: Influence of Edible Marijuana on Endurance Exercise Performance
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Christopher Bell (Other)
Responsible Party: Sponsor-Investigator, Christopher Bell, Associate Professor, Colorado State University
Organization: Colorado State University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2827
Record Dates: First submitted 2021-12-31; First posted 2022-01-14 (Actual); Results first posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Endurance Exercise
MeSH Terms: interventions — THC 5

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either placebo or intervention separated by a 4 day wash-out period.
Who Masked: Participant
Masking Description: Coded envelope.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Delta-9-tetrahydrocannabinol (THC) free fruit snack gummy. One time, two gummies will be ingested prior to an exercise bout.
  Interventions: Drug: Placebo
- 10 mg THC (Active Comparator): Delta-9-tetrahydrocannabinol (THC) 5 milligrams (mg) in gummy form. One time, two gummies will be ingested prior to an exercise bout.
  Interventions: Drug: THC 5

INTERVENTIONS:
Drug: THC 5 — 5 milligrams of THC in gummy form
  Other Names: Ripple Blood Orange Gummies (Stillwater Brands, Commerce City, CO).
  Arms: 10 mg THC
Drug: Placebo — Commercially available non-THC fruit snack
  Other Names: Welch Fruit Snack
  Arms: Placebo

SUMMARY:
Lots of people, including athletes and people who like to exercise regularly, enjoy marijuana. Some people believe marijuana might improve their ability to exercise. There are no recent, up-to-date scientific studies to suggest that this belief is right or wrong. The goal of this study is to determine the influence of marijuana on exercise performance.

DETAILED DESCRIPTION:
The purpose of the proposed project is to provide athletes and the scientific community with data pertaining to the acute influence of edible marijuana on exercise performance, and the physiological responses to standardized exercise. Specifically, the investigators wish to determine: 1. The influence of edible marijuana on cardio-respiratory and metabolic responses to standardized cycle ergometer exercise. 2. The influence of edible marijuana on endurance exercise (time-trial) performance.

The investigators wish to determine if edible marijuana, ingested prior to exercise, is ergogenic (improves performance) or ergolytic (decreases performance).

The investigators hypothesize that edible marijuana will be ergolytic.

ELIGIBILITY:
Inclusion Criteria:

* Between the age of 21 and 40.
* Weigh more than 110 pounds
* Habitual user of cannabis; average use of THC minimum of once per month during the previous year
* Prior use of cannabis product containing at least 10 mg of THC with no adverse reaction
* Habitual exerciser: exercised a minimum of 5 days per week, for a minimum of 30-minutes/session, during the previous year.

Exclusion Criteria:

* Identification of a contra-indication to exercise during a 12-lead exercise stress test.
* Pregnant or trying to become pregnant. Breastfeeding.
* Recipient of treatment for psychotic or bipolar disorder during the previous 2 years
* Recipient of treatment for Schizophrenia during the previous 2 years
* Planned surgery scheduled within 2-weeks of study participation

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2022-07-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Colorado State University, Dept. of Health and Exercise Science, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to Published Manuscript — https://pubmed.ncbi.nlm.nih.gov/36545283/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Seventeen adults were assessed for eligibility and enrolled in the study. Two adults declined invitations to schedule post-screening study visits, two were excluded from participation on account of use of contraindicated medications, and three were discontinued during the habituation visits as they were unable to sustain the required work rate. This all occurred prior to treatment assignments (randomization).
Groups:
- THC Gummy First, Then Placebo Gummy: Delta-9-tetrahydrocannabinol (THC) 5 milligrams (mg) in gummy form. One time, two gummies will be ingested prior to an exercise bout.
  THC 5: 5 milligrams of THC in gummy form
  4-day minimum washout period
  Delta-9-tetrahydrocannabinol (THC) free fruit snack gummy. One time, two gummies will be ingested prior to an exercise bout.
  Placebo: Commercially available non-THC fruit snack
- Placebo Gummy First, Then THC Gummy: Delta-9-tetrahydrocannabinol (THC) free fruit snack gummy. One time, two gummies will be ingested prior to an exercise bout.
  Placebo: Commercially available non-THC fruit snack
  4-day minimum washout period
  Delta-9-tetrahydrocannabinol (THC) 5 milligrams (mg) in gummy form. One time, two gummies will be ingested prior to an exercise bout.
  THC 5: 5 milligrams of THC in gummy form
Period: Overall Study
Arm/Group | THC Gummy First, Then Placebo Gummy | Placebo Gummy First, Then THC Gummy
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 10 participants completed both measures (Placebo and THC). 9 participants were analyzed. 1 participant was excluded from analyses due to failure to abstain.
Groups:
- Randomized Crossover Study: Participants first received either a Placebo gummy (commercially available non-THC fruit snack) or 2 5mg THC gummies prior to an exercise bout. Visits were separated by a 4-day washout period.
Arm/Group | Randomized Crossover Study
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height [Mean (Standard Deviation); unit: cm] | 167.3 (25.5)
Body Mass [Mean (Standard Deviation); unit: kg] | 75.97 (13.30)
Lean Mass [Mean (Standard Deviation); unit: kg] | 57.98 (9.79)
Body Fat [Mean (Standard Deviation); unit: % of body fat] | 20.12 (3.05)
VO2 peak [Mean (Standard Deviation); unit: L/min] — Peak oxygen uptake
  L/min | 4.34 (1.26)
VO2 peak [Mean (Standard Deviation); unit: ml/kg/min] — Peak oxygen uptake.
  ml/kg/min | 56.5 (11.7)

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Blood Lactate Levels During a 24 Minute Graded Standard Exercise Test (50 Watts, 100 Watts, and 150 Watts) to Placebo.
Description: Separated by a minimum of a 4 day washout period between randomized crossover coded interventions. Blood will be collected to determine Blood Lactate Levels during standard exercise following ingestion of placebo or active formula.
Time Frame: Blood was collected at timepoints 0 minutes (0 watts), 8 minutes (50 watts), 16 minutes (100 watts), and 24 minutes (150 watts) for analysis of blood lactate.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Placebo | 10 mg THC
Number analyzed (Participants) | 9 | 9
mmol/L
  0 minutes - 0 watts | 0.9699 (0.3711208) | 1.1437 (0.358376)
  8 minutes - 50 watts | 1.26345 (0.47071) | 1.3618 (0.343596)
  16 minutes - 100 watts | 1.6075 (0.9670983) | 1.3558333 (0.7374943)
  24 minutes - 150 watts | 2.5896 (2.254174) | 2.4418 (2.2780711)

2. Primary Outcome: Comparison of Heart Rate During a 24 Minute Graded Standard Exercise Test (50 Watts, 100 Watts, and 150 Watts) to Placebo.
Description: Separated by a minimum of a 4 day washout period between randomized crossover coded interventions.Heart rate will be collected during standard graded exercise following ingestion of placebo or active formula (10mg THC in the form of two 5mg gummies).
Time Frame: Heart rate was measured at timepoints 0 minutes (0 watts), 8 minutes (50 watts), 16 minutes (100 watts) and 24 minutes (150 watts)
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Placebo | 10 mg THC
Number analyzed (Participants) | 9 | 9
bpm
  0 minutes - 0 watts | 66 (16) | 63 (13)
  8 minutes - 50 watts | 95 (14) | 97 (15)
  16 minutes - 100 watts | 108 (18) | 113 (20)
  24 minutes - 150 watts | 130 (26) | 135 (27)

3. Primary Outcome: Comparison of Rating of Perceived Exertion (RPE) During a 24 Minute Graded Standard Exercise Test (50 Watts, 100 Watts, and 150 Watts) to Placebo.
Description: Separated by a minimum of a 4 day washout period between randomized crossover coded interventions.During standard exercise, participants will be asked to report Rating of Perceived Exertion (RPE) on a scale from 6-20 (6 is no exertion and 20 is maximal exertion) during a graded standard exercise test following ingestion of placebo or active formula.
Time Frame: RPE was reported and averaged for each intensity stage at timepoints 0 minutes- 4 minutes (0 watts), 8 minutes-12 minutes (50 watts), 16 minutes-20 minutes (100 watts), and 24 minutes (150 watts).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | 10 mg THC
Number analyzed (Participants) | 9 | 9
units on a scale
  0 and 4 minutes - 0 watts | 6 (0) | 6 (0)
  8 and 12 minutes - 50 watts | 8 (1) | 8 (1)
  16 and 20 minutes - 100 watts | 11 (1) | 10 (1)
  24 minutes - 150 watts | 12 (1) | 12 (1)

4. Primary Outcome: Comparison of Indirect Calorimetry (VO2) During a 24 Minute Graded Standard Exercise Test (50 Watts, 100 Watts, and 150 Watts) to Placebo.
Description: Separated by a minimum of a 4 day washout period between randomized crossover coded interventionsVO2 will be collected during graded standard exercise following ingestion of placebo or active formula. Expired gasses were measured and averaged during three time points, 5-8 minutes, 13-16 minutes, and 21-24 minutes. Gasses were not collected or recorded outside of those timeframes.
Time Frame: Expired gasses were measured and averaged during three time points, 5-8 minutes (50 Watts), 13-16 minutes (150 Watts), and 21-24 minutes (150 Watts).
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Placebo | 10 mg THC
Number analyzed (Participants) | 9 | 9
L/min
  5-8 minutes- 50 watts | 1.26404 (0.31999) | 1.24939816 (0.15584784)
  13-16 minutes-100 watts | 1.66361 (0.18041) | 1.664867728 (0.138618921)
  21-24 minutes- 150 watts | 2.11388 (0.15106) | 2.126941406 (0.133666814)

5. Primary Outcome: Comparison of Maximal Mean Power Output to Placebo
Description: Mean maximal power will be measured over 20 minutes following ingestion of placebo or active formula
Time Frame: Separated by a minimum of a 4 day washout period between randomized crossover coded interventions
Measure: Mean (Standard Deviation); unit: watts
Arm/Group | Placebo | 10 mg THC
Number analyzed (Participants) | 9 | 9
watts | 422 (92) | 454 (77)

6. Primary Outcome: Comparison of Time to Exhaustion to Placebo
Description: Cycling until Time to Exhaustion in seconds following ingestion of placebo or active formula during high intensity exercise
Time Frame: Separated by a minimum of a 4 day washout period between randomized crossover coded interventions.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Placebo | 10 mg THC
Number analyzed (Participants) | 9 | 9
seconds | 43 (33) | 43 (32)

ADVERSE EVENTS:
Time Frame: Each study participant was monitored for Adverse Events for 30 minutes post-invention, with a 4-day washout period in between interventions. During the 24 hours post-intervention, study participants were instructed to email study staff to report new or recurring events.
Arm/Group | Placebo | 10 mg THC
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-12-31): https://cdn.clinicaltrials.gov/large-docs/39/NCT05192239/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-05): https://cdn.clinicaltrials.gov/large-docs/39/NCT05192239/SAP_001.pdf
  • Informed Consent Form (2021-10-27): https://cdn.clinicaltrials.gov/large-docs/39/NCT05192239/ICF_002.pdf